CLINICAL TRIAL: NCT04642664
Title: Apatinib Plus Camrelizumab in Patients With Previously Treated Advanced Biliary Tract Cancer (ACABC): A Prospective Clinical Study
Brief Title: Apatinib Plus Camrelizumab in Patients With Previously Treated Advanced Biliary Tract Cancer
Acronym: ACABC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-2160
Record Dates: First submitted 2020-11-22; First posted 2020-11-24 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2020-11

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma; Biomarker; Hepatobiliary Neoplasm
Keywords: apatinib; camrelizumab; biliary tract cancer; combination immunotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — apatinib; camrelizumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib plus Camrelizumab (Experimental): Apatinib is a multi-target TKI, which selectively inhibits VEGFR-2.
  Camrelizumabb is a anti-human PD-1 monoclonal antibody.
  Interventions: Drug: Apatinib plus Camrelizumab

INTERVENTIONS:
Drug: Apatinib plus Camrelizumab — Patients received apatinib orally at 250 mg once a day irrespective of the patient weight. During the treatment, apatinib can reduced to half of piece or once every other day considering the grade of treatment related adverse events. Camrelizumab 200 mg was administered intravenously over 30 minutes every 3 weeks. The intermittent period of camrelizumab was no longer than 6 weeks. All patients continued combination treatment until disease progression, unacceptable toxicity, or discontinuation for any reason.
  Other Names: Apatinib (Apatinib Mesylate Tablets, Jiangsu Hengrui Medicine, China); Camrelizumab (Carelizumab for Injection, Jiangsu Hengrui Medicine, China)

SUMMARY:
The investigators design a prospective clinical study to explore the efficacy and safety of apatinib plus camrelizumab in pretreated patients with advanced biliary tract malignant tumors and to analyze potential biomarkers of therapeutic response.

DETAILED DESCRIPTION:
This was a non-randomized, single institutional, open-label, prospective trial designed to evaluate the efficacy and safety of apatinib in combination with camrelizumab for patients with biliary tract malignant tumors.

It is estimated that 20 patients who met the study criteria will be enrolled in PUMCH and treated with aptinib and camrelizumab. The investigators will follow up and collect subjects' data each month to evaluate the efficacy and safety of treatment, including treatment related adverse events, overall survival and time to progression and objective response. Multi-omics data analysis will be used to find potential biomarkers of treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed cholangiocarcinoma including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma and gallbladder cancer. Patients with ampullary carcinoma are not eligible.
2. Patients must have failed or are intolerant to one line of systemic chemotherapy treatment.
3. Patients who received adjuvant chemotherapy and had evidence of disease recurrence within 6 months of completion of the adjuvant treatment are also eligible. If the patient received adjuvant treatment and had disease recurrence after 6 months, patients will only be eligible after failing or having intolerance to one line of systemic chemotherapy used to treat the disease recurrence.
4. Age ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status Assessment of 0-2.
6. Life expectancy of at least 12 weeks (3 months).
7. Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other study requirements.
8. All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v4.0 Grade 1 or less at the time of signing the Informed Consent Form (ICF) except for alopecia.
9. For patients with advanced biliary tract cancer, liver function status Child-Pugh Class A or B (score<=7).
10. Adequate bone marrow, liver and liver function as assessed by the following laboratory requirements: Total bilirubin ≤ 1.5 x the upper limits of normal (ULN), except for subjects with Gilbert Syndrome who can have bilirubin <3. Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer or stent placement). Alkaline phosphastase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer). Serum creatinine <2 x ULN. Hematologic parameters as follows: Platelet count ≥ 100,000 /mm3. Hemoglobin (Hb) ≥ 9 g/Dl. Absolute neutrophil count (ANC) ≥1000/mm. Blood transfusion to meet the inclusion criteria will be allowed.
11. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity of 25 IU/L or equivalent units of HCG) performed within24 hours prior to the start of nivolumab Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
12. Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 3 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
13. Patients with history of hepatitis B and hepatitis C will be eligible but patients with hepatitis B must be started on antiviral therapy prior to beginning study therapy
14. Availability of archival tumor tissue for biomarkers analysis (FFPE block or cell block will be required). Specimen from primary site will be allowed. Patients must have at least 10 slides available. Repeat biopsy to obtain sufficient tissue for 10 slides is allowed.

Exclusion Criteria

1. Subjects with active CNS metastases are excluded. If CNS metastases are treated and subjects are at neurologic baseline for at least 2 weeks prior to enrollment, they will be eligible but will need a Brain MRI prior to enrollment. Subjects must be off corticosteroids or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).
2. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
3. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
4. Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
5. Known history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
6. Child Pugh C disease
7. History of severe hypersensitivity reactions to other monoclonal antibodies
8. History of allergy or intolerance to study drug components or Polysorbate-80-containing infusions
9. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
10. History or concurrent condition of interstitial lung disease of any grade or severely impaired pulmonary function.
11. Unresolved toxicity higher than CTCAE grade 1 attributed to any prior therapy/procedure excluding alopecia.
12. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity of 25 IU/L or equivalent units of HCG) performed within 24 hours prior to the start of nivolumab and a negative result must be documented before start of treatment.
13. Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his/her compliance in the study.
14. Anticancer chemotherapy during the study or within 4 weeks of study enrollment. Subjects must have recovered from the toxic effects of the previous anti-cancer chemotherapy (with the exception of alopecia). Anti-cancer therapy is defined as any agent or combination of agents with clinically proven anti-tumor activity administered by any route with the purpose of affecting the malignancy, either directly or indirectly, including palliative and therapeutic endpoints.
15. Hormonal therapy during the study or within 2 weeks of first study enrollment.
16. Investigational drug therapy outside of this trial during or within 4 weeks of first study treatment.
17. Notably, patients with severe esophageal varices or presented with positive fecal occult blood were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Six months
  A duration from the date of initial treatment with apatinib plus camrelizumab to disease progression (defined by RECIST 1.1) or death of any cause.
Objective Response Rate (ORR) | One year
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.

SECONDARY OUTCOMES:
Overall Survival (OS) | Two years
  Duration from the date of initial treatment with apatinib plus camrelizumab to the date of death due to any cause
Incidence of Treatment-Emergent Adverse Event | Two years
  Any adverse events related with treatment with apatinib plus camrelizumab

OTHER OUTCOMES:
Clinical benefit rate (CBR) | Six months
  The CBR was defined as the proportion of patients who achieved a radiologically confirmed objective response (CR or PR) or who had PFS time longer than 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Tao Zhao, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Chinese Academy of Medical Sciences & Peking Union Medical College Hospital (CAMS&PUMCH), Beijing, Beijing Municipality
  - Hai-Tao Zhao, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Razumilava N, Gores GJ. Cholangiocarcinoma. Lancet. 2014 Jun 21;383(9935):2168-79. doi: 10.1016/S0140-6736(13)61903-0. Epub 2014 Feb 26. PMID 24581682
- [Result] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Result] Scott LJ. Apatinib: A Review in Advanced Gastric Cancer and Other Advanced Cancers. Drugs. 2018 May;78(7):747-758. doi: 10.1007/s40265-018-0903-9. PMID 29663291
- [Result] Hu Y, Lin H, Hao M, Zhou Y, Chen Q, Chen Z. Efficacy and Safety of Apatinib in Treatment of Unresectable Intrahepatic Cholangiocarcinoma: An Observational Study. Cancer Manag Res. 2020 Jul 3;12:5345-5351. doi: 10.2147/CMAR.S254955. eCollection 2020. PMID 32753952
- [Result] Xu J, Shen J, Gu S, Zhang Y, Wu L, Wu J, Shao G, Zhang Y, Xu L, Yin T, Liu J, Ren Z, Xiong J, Mao X, Zhang L, Yang J, Li L, Chen X, Wang Z, Gu K, Chen X, Pan Z, Ma K, Zhou X, Yu Z, Li E, Yin G, Zhang X, Wang S, Wang Q. Camrelizumab in Combination with Apatinib in Patients with Advanced Hepatocellular Carcinoma (RESCUE): A Nonrandomized, Open-label, Phase II Trial. Clin Cancer Res. 2021 Feb 15;27(4):1003-1011. doi: 10.1158/1078-0432.CCR-20-2571. Epub 2020 Oct 21. PMID 33087333
- [Result] Liu J, Liu Q, Li Y, Li Q, Su F, Yao H, Su S, Wang Q, Jin L, Wang Y, Lau WY, Jiang Z, Song E. Efficacy and safety of camrelizumab combined with apatinib in advanced triple-negative breast cancer: an open-label phase II trial. J Immunother Cancer. 2020 May;8(1):e000696. doi: 10.1136/jitc-2020-000696. PMID 32448804
- [Result] Liang L, Wen Y, Hu R, Wang L, Xia Y, Hu C, Qiao Y, Geng X, Chen T, Fei J, Hui K, Jiang X. Safety and efficacy of PD-1 blockade-activated multiple antigen-specific cellular therapy alone or in combination with apatinib in patients with advanced solid tumors: a pooled analysis of two prospective trials. Cancer Immunol Immunother. 2019 Sep;68(9):1467-1477. doi: 10.1007/s00262-019-02375-z. Epub 2019 Aug 27. PMID 31451841
- [Result] Xie L, Xu J, Sun X, Guo W, Gu J, Liu K, Zheng B, Ren T, Huang Y, Tang X, Yan T, Yang R, Sun K, Shen D, Li Y. Apatinib plus camrelizumab (anti-PD1 therapy, SHR-1210) for advanced osteosarcoma (APFAO) progressing after chemotherapy: a single-arm, open-label, phase 2 trial. J Immunother Cancer. 2020 May;8(1):e000798. doi: 10.1136/jitc-2020-000798. PMID 32376724
- [Result] Franses JW, Hong TS, Zhu AX. Nivolumab with gemcitabine plus cisplatin for biliary cancers: as easy as ABC? Lancet Gastroenterol Hepatol. 2019 Aug;4(8):575-577. doi: 10.1016/S2468-1253(19)30148-7. Epub 2019 May 17. No abstract available. PMID 31109809
- [Result] Qin S, Ren Z, Meng Z, Chen Z, Chai X, Xiong J, Bai Y, Yang L, Zhu H, Fang W, Lin X, Chen X, Li E, Wang L, Chen C, Zou J. Camrelizumab in patients with previously treated advanced hepatocellular carcinoma: a multicentre, open-label, parallel-group, randomised, phase 2 trial. Lancet Oncol. 2020 Apr;21(4):571-580. doi: 10.1016/S1470-2045(20)30011-5. Epub 2020 Feb 26. PMID 32112738
- [Derived] Wang D, Yang X, Long J, Lin J, Mao J, Xie F, Wang Y, Wang Y, Xun Z, Bai Y, Yang X, Guan M, Pan J, Seery S, Sang X, Zhao H. The Efficacy and Safety of Apatinib Plus Camrelizumab in Patients With Previously Treated Advanced Biliary Tract Cancer: A Prospective Clinical Study. Front Oncol. 2021 Apr 12;11:646979. doi: 10.3389/fonc.2021.646979. eCollection 2021. PMID 33912461